CLINICAL TRIAL: NCT00526448
Title: Open, Multicentre,Randomized Phase IV Trial to Evaluate Efficacy/Safety to Extend Treatment Duration With Peginterferon Alfa-2a+High Dose of Ribavirin Supporting Epo β in Treatment of CHC in HIV-HCV Patients Who Not Clear Virus at Week 4
Brief Title: Phase IV Study to Evaluate the Efficacy/Safety to Extend Treatment and High Dose of Ribavirin in co-Infected Patients
Acronym: PERICO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Carlos III, Madrid (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-005940-99
Record Dates: First submitted 2007-09-05; First posted 2007-09-10 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Chronic Hepatitis C
Keywords: high dose of ribavirin; extend treatment duration; tailoring treatment
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2a; epoetin beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Peginterferon alfa-2a 180 mcg/week + ribavirin 2000 mg/day + epoetin beta 450 UI/week
  Interventions: Drug: ribavirin; Drug: Peginterferon alfa-2a; Drug: epoetin beta
- 2 (Active Comparator): Peginterferon alfa-2a 180 mcg/week + ribavirin 1000-1200 mg/day
  Interventions: Drug: ribavirin; Drug: Peginterferon alfa-2a

INTERVENTIONS:
Drug: ribavirin — 2000 mg/day
  Arms: 1
Drug: ribavirin — 1000-1200 mg/day
  Arms: 2
Drug: Peginterferon alfa-2a — Peginterferon alfa-2a 180 mcg/week
Drug: epoetin beta — epoetin beta 450 UI/week
  Arms: 1

SUMMARY:
To compare the sustained virological response (SVR = ribonucleic acid (RNA) - hepatitis C virus (HCV) undetectable at week 24 before end the treatment) in chronic hepatitis C patients genotype 1-4 co-infected with HIV-HCV, treated with Peginterferón alfa-2a (40 KD) 180 µg/week and Ribavirin (2000 mg/day during 4 weeks, follow of 1000-1200 mg/day, according to body weight); versus Peginterferón alfa-2a (40 KD) 180 μg/week and Ribavirin (1000-1200 mg/day, according to body weight).

To evaluate the impact to extend the treatment with Peginterferon alfa-2a and Ribavirin to week 72, in SVR of these patients with genotypes 1-4 without rapid virological response (RVR = RNA - HCV undetectable at 4 week).

DETAILED DESCRIPTION:
The PRESCO study (ribavirin dose 1000-1200 mg/day) emphasized that optimal ribavirin exposure seems to be crucial to maximize sustained virological response and minimize the incidence of relapses after treatment discontinuations.

Recent reports showed that it is beneficial to extend the treatment duration in patients without rapid virological response at 4 weeks (RNA-HCV < 50 UI/ml).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients > 18 years of age
* Serologic evidence of anti-HCV
* Detectable plasma HCV-RNA
* Serologic evidence of HIV-1 infection
* CD4 cell count >/= 250 cell/mm3
* Stable status of HIV-1 infection in the opinion of the investigator
* Patients on stable antiretroviral therapy (HAART) for at least 6 weeks prior to baseline whose HAART regimen (drugs and dosage) is expected to remain unaltered for the first 6 weeks of this study
* Patients who have not been on HAART for at least 6 weeks prior to randomization who are willing to delay initiation of HAART therapy for at least 6 weeks
* Negative urine or blood pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of study drug
* Willingness to give written informed consent

Exclusion Criteria:

* Women with ongoing pregnancy or breast feeding
* Male partners of women who are pregnant
* IFN/ribavirin therapy at any previous time
* Child Pugh > 6 (Child Pugh B or C)
* History or conditions consistent with decompensated liver disease
* Any investigational drug 6 weeks prior to the first dose of study drug (expanded access programs for HIV treatment are allowed)
* Patients treated with didanosine and/or zidovudine
* Positive test at anti-HAV IgM Ab, HBsAg, anti-HBc IgM Ab, HBeAg
* History or other evidence of a medical condition associated with chronic liver disease other than HCV
* Hepatocarcinoma observed in the liver ecography
* Serum concentrations of ceruloplasmin or alfa1-antitrypsin at screening consistent with an increased risk of metabolic liver disease
* Active HIV-related opportunistic infection and/or malignancy requiring acute systemic therapy
* Absolute neutrophil count (ANC) < 1500 cells/mm3
* Hgb < 11 g/dL in women or 12 g/dL in men or any patient for whom anemia would be medically problematic
* Hemoglobinopathy or any other cause of or tendency for hemolysis
* Platelet count < 50,000 cells/mm3
* History of G-CSF, GM-CSF or epo treatment during 3 months prior to the first dose of study drug
* Serum creatinine level > 1.5 times the upper limit of normal at screening
* History of severe psychiatric disease, especially depression
* History of a severe seizure disorder or current anticonvulsant use
* History of immunologically mediated disease
* History or other evidence of chronic pulmonary disease associated with functional limitation
* History of significant cardiac disease that could be worsened by acute anemia
* History of thyroid disease poorly controlled on prescribed medications
* Evidence of severe retinopathy
* History of major organ transplantation with an existing functional graft
* History or other evidence of severe illness, malignancy or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
* History of any systemic anti-neoplastic or immunomodulatory treatment 6 months prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study
* Concomitant medication with rifampin/rifampicin, rifabutin, pyrazinamide, isoniazid, gancyclovir, thalidomide, oxymetholone, immunomodulatory treatments and systemic antiviral agents as adjuvant therapy for CHC
* Drug use within 6 months of 1st dose and excessive alcohol consumption

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2007-06; Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
% patients with RNA-HCV < 50 UI/ml | 24 weeks after the end of treatment

SECONDARY OUTCOMES:
% patients with RNA-HCV < 50 UI/ml | 4 weeks on treatment

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Soriano, Dr, Study Chair — Hospital Carlos III. Madrid. Spain
Locations (40):
- Spain (40):
  - Hospital Juan Canalejo, A Coruña, A Coruña
  - Hospital Txagorritxu, Vitoria-Gasteiz, Alava
  - Hospital de Albacete, Albacete, Albacete
  - Hospital General de Elche, Elche, Alicante
  - Hospital Son Dureta, Palma de Mallorca, Balearic Islands
  - Hospital Santa Creu y Sant Pau, Barcelona, Barcelona
  - Hospital Parc Taulí, Sabadell, Barcelona
  - Hospital General de Jerez de la Frontera, Jerez de la Frontera, Cadiz
  - Hospital Marqués de Valdecilla, Santander, Cantabria
  - Hospital General de Fuerteventura, Puerto del Rosario, Fuerteventura
  - Hospital Doctor Negrín, Las Palmas de Gran Canarias, Gran Canaria
  - Hospital Clínico san Cecilio, Granada, Granada
  - Hospital San Jorge, Huesca, Huesca
  - Hospital Arquitecto Marcide, Ferrol, La Coruña
  - Hospital Clínico Universitario, Santiago, La Coruña
  - Hospital Xeral-Caldé, Lugo, Lugo
  - Hospital de Alcorcon, Alcorcón, Madrid
  - Hospital Severo Ochoa, Leganés, Madrid
  - Hospital de la Princesa, Madrid, Madrid
  - Hospital Gregorio Marañón, Madrid, Madrid
  - Hospital Carlos III, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital Santa Maria del Rosell, Murcia, Murcia
  - Hospital Clínico Virgen de la Victoria, Málaga, Málaga
  - Hospital Xeral-Cíes, Vigo, Pontevedra
  - Hospital do Meixoeiro, Vigo, Pontevedra
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Clínico de Salamanca, Salamanca, Salamanca
  - Hospital General de la Palma, La Palma, Santa Cruz de Tenerife
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz de Tenerife
  - Hospital de la Candelaria, Santa Cruz de Tenerife, Santa Cruz de Tenerife
  - Hospital Virgen de la Macarena, Seville, Sevilla
  - Hospital de Valme, Seville, Sevilla
  - Hospital Universitario la Fé, Valencia, Valencia
  - Hospial Clinico Universitario de Valencia, Valencia, Valencia
  - Hospital Clínico de Valladolid, Valladolid, Valladolid
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza, Zaragoza
  - Hospital Miguel Servet, Zaragoza, Zaragoza

REFERENCES:
- [Derived] Vispo E, Labarga P, Guardiola JM, Barreiro P, Miralles C, Rubio R, Miralles P, Aguirrebengoa K, Portu J, Morello J, Rodriguez-Novoa S, Soriano V; PERICO Study Group. Preemptive erythropoietin plus high ribavirin doses to increase rapid virological responses in HIV patients treated for chronic hepatitis C. AIDS Res Hum Retroviruses. 2010 Apr;26(4):419-24. doi: 10.1089/aid.2009.0120. PMID 20377423